CLINICAL TRIAL: NCT03304600
Title: Transcranial Direct Current Stimulation (tDCS) to Treat Patients With Severe and Resistant Obsessive Compulsive Disorder
Brief Title: tDCS for Treatment Resistant Obsessive Compulsive Disorder
Acronym: tDCS-TOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-A01983-48
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; tDCS
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): 10 sessions (1 per day during 2 week) of active tDCS stimulation
  Interventions: Device: Active stimulation
- Sham Stimulation (Sham Comparator): 10 sessions (1 per day during 2 week) of sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Active stimulation — Patients will receive a tDCS stimulation during 30 mn with an intensity of 2 milliampere (mA).
  Arms: Active stimulation
Device: Sham stimulation — Patients will receive a Sham stimulation during 30 mn
  Arms: Sham Stimulation

SUMMARY:
It's a multicentric, randomized, controlled study concerning 100 patients with treatment-resistant obsessive compulsive disorders (OCD). The aim of this study is to evaluate the effect of transcranial direct current stimulation (tDCS) on OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for obsessive compulsive disorder according to Diagnostic and Statistical Manual (DSM IV) with a "good insight" (BABS)
* No current depressive and suicidal risks
* No epileptic pathology
* Age: Participants will be both males and females, 18-70 years of age included.
* Chronic Obsessive compulsive disorder ( Total Y-BOCS>20 or Y-BOCS one subscale > 15)
* Obsessive compulsive disorder resistant to pharmacology treatment :

  1. at least 2 antidepressants (IRS type) (> 12 weeks)
  2. cognitive and comportment therapy since at least one year
* Treatment stability (antidepressants) for more than 12 weeks without significant improvement.
* Affiliation to a social security system (recipient or assignee),
* Signed written inform consent form

Exclusion Criteria:

* Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception or who is nursing,
* Patient under curators
* Patient hospitalized under duress
* Meets another diagnosis of axe 1 of DSM-IV
* Current depressive or suicidal risks
* Patient with any form of metal in the cranium, a pacemaker, skull defects, or skin lesions to the scalp (cuts, abrasions, rash)
* Epileptic patient
* Patient with a medical history of cranial trauma
* Patient unable to give his or hers informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) score | 2 weeks
  The primary objective of the study is to compare the change in Yale Brown Obsessive Compulsive Scale (YBOCS) scores from baseline to the week 2 (post-tDCS treatment) visit, between the two treatments groups

SECONDARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale (YBOCS) | Month 1
  i. Change from baseline to month 1 in Yale Brown Obsessive Compulsive Scale (YBOCS) scores, between treatment groups.
Yale Brown Obsessive Compulsive Scale (YBOCS), | Month 3
  ii. Response rate at month 3 in Yale Brown Obsessive Compulsive Scale (YBOCS) score from baseline, between treatment groups.
Clinical Global Impression (CGI) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Clinical Global Impression (CGI) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;
Brown Assessment of Beliefs Scale (BABS) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Brown Assessment of Beliefs Scale (BABS) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;
Brief Anxiety Scale (BAS) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Brief Anxiety Scale (BAS) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;
Montgomery and Asberg Depression Rating Scale (MADRS) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Montgomery and Asberg Depression Rating Scale (MADRS) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;
Hospital Anxiety and Depression scale (HAD) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Hospital Anxiety and Depression scale (HAD) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;
Sheehan Disability Scale, (SDS) | Month 1
  Change from baseline to month 1 in above scales between treatment groups;
Sheehan Disability Scale, (SDS) | Month 3
  Change from baseline to month 3 in above scales between treatment groups;

OTHER OUTCOMES:
Number of adverse events | 3 Month
  Safety of the tDCS treatment :
  * assessed by physical examination during each tDCS session
  * any other adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Damien HEIT, MD, Study Director — Centre Hospitalier Henri Laborit
Locations (4):
- France (4):
  - Hospices Civils De Lyon, Lyon
  - CHU de Nantes, Nantes
  - Centre Hospitalier Henri Laborit, Poitiers
  - C.H. Guillaume Regnier, Rennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harika-Germaneau G, Heit D, Drapier D, Sauvaget A, Bation R, Chatard A, Doolub D, Wassouf I, Langbour N, Jaafari N. Treating refractory obsessive compulsive disorder with cathodal transcranial direct current stimulation over the supplementary motor area: a large multisite randomized sham-controlled double-blind study. Front Psychiatry. 2024 May 17;15:1338594. doi: 10.3389/fpsyt.2024.1338594. eCollection 2024. PMID 38827437